CLINICAL TRIAL: NCT05430139
Title: Dried Blood Spot Testing for At Home Health
Status: Recruiting | Type: Observational
Sponsor: Switch Health Solutions Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DBS-01
Record Dates: First submitted 2022-06-15; First posted 2022-06-24 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Diabetes; Thyroid Diseases
MeSH Terms: conditions — Diabetes Mellitus; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DBS (Dried blood spot) is the collection of a small volume of blood on paper cards and subsequent transport to an analytical laboratory. This method is widely used for newborn screening programs around the world to identify inborn errors of metabolism where early diagnosis and treatment can be lifesaving. The World Health Organization and World Anti-Doping Agency (WADA) have independently endorsed DBS as an alternative to conventional testing methods due to its lessened invasiveness, lower collection and transport cost, reduction in sample storage needs, and for some analytes, improved sample stability. There are hundreds of publications describing DBS testing and some commercial ventures offering direct-to-consumer testing using DBS. However, it is not clear if there have been concerted efforts to develop DBS sampling for adults for home collection in concert with high quality, accredited central clinical laboratories. The proposal herein is focused on developing and validating DBS for at home and remote sample collections for routine diagnostic testing.

DETAILED DESCRIPTION:
Remote phlebotomy services have long been an option for remote communities, yet through the pandemic there has been an apparent decline in these facilities likely driven by a lack of financial incentive for community laboratories; outpatient test volumes decreased in the early months of the pandemic and cuts commensurate with these revenue losses either reduced access or pushed the work to hospital laboratories. Sample stability and transportation for remote sites is also challenging and expensive.

Point of care (POC) testing options are an area of active research and development (R&D) and are generally attractive for healthcare providers and patients. However, POC testing does suffer in terms of quality and accuracy, even in the hands of trained nursing professionals. Preanalytical errors, problems that occur with sample collection, device quality control and storage, still plague POC testing. In addition, POC tests tend to be more expensive than central laboratory tests and there is an underappreciation of the skill required to perform tests accuracy.

Remote self-sample collection and transport to central labs for analysis has several options, the most promising of which is dried blood spot (DBS) testing. DBS is the collection of a small volume of blood on paper cards. DBS samples are largely stable and may be collected at home or outside of the usual healthcare facilities and transported to a clinical laboratory for analysis. This method is widely used for newborn screening programs around the world to identify inborn errors of metabolism where early diagnosis and treatment can be lifesaving. The World Health Organization has also endorsed DBS for testing for human immunodeficiency virus (HIV) and hepatitis B and C infection in remote and hard to reach populations. The WHO states that DBS samples are effective for measuring antibodies, serologic antigens, and nucleic acids using commonly available commercial laboratory methods. Recently the World Anti-Doping Agency (WADA) endorsed DBS testing for performance enhancing drugs. WADA cites benefits of easy sample collection, less invasive methods than current observed urine and blood collection and therefore, less expensive collection and transport of samples, reduction in sample storage needs, and for some analytes, improved sample stability.

There are hundreds of publications describing DBS testing and some commercial ventures offering direct-to-consumer testing using DBS. However, it is not clear if there have been concerted efforts to develop DBS sampling for adults for home collection in concert with high quality, accredited central clinical laboratories. This partly stems from the additional effort and cost needed to process DBS samples and the need for extensive validation studies to ensure robustness, accuracy, and precision. The proposal herein is focused on developing and validating DBS for at home and remote sample collections for routine diagnostic testing.

ELIGIBILITY:
Inclusion Criteria:

1. Participant >=18 years old.
2. Visiting Bio-Test Laboratory for routine, physician-ordered venous blood collection.
3. Able to provide informed consent.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent.
2. Pre-existing coagulopathies that might put them at risk for bleeding (e.g., hemophilia)
3. Unable to produce an adequate blood sample.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include 2000 participants who will be recruited when visiting Bio-Test Laboratory for routine, physician-ordered bloodwork (venous blood collection).
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Method Comparison Studies | Through study completion - approximately 6 months
  For comparisons, routine commercial diagnostic methods will be used as the predicate. The gold standard will be defined as antecubital vein venous blood collections into lithium heparin with gel separator (or serum separator tubes) for thyroid hormones, and K2-EDTA tubes for HbA1c analysis. Any commercially available clinical valid method performed in an accredited laboratory would serve as an acceptable reference method. Comparison studies will require 200 samples spanning the analytical measuring range of the assay. Paired venous collections will be required for comparison.
Precision Studies | Through study completion - approximately 6 months
  Precisions studies will be performed first using CLSI EP05A3 recommendations for within run, within day, between day, and total imprecision using commercial controls. This routine analysis will be augmented with repeat analysis of DBS samples to assess the stability of the matrix and the ability to extract analytes reproducibly. To assess reproducibility in patient samples, 20 sets of samples (of varying concentration) will be tested in triplicate on serial days (3x5).
Linearity Studies | Through study completion - approximately 6 months
  Linearity studies will be performed using known standards (e.g. NIST, assayed controls, EQA material) diluted to challenge the vendor claim. Where necessary, dilutions will be done according to the vendor instructions for users. CLSI EP06 (Evaluation of Linearity) will be followed using triple samples fit with sequential polynomials (1st, 2nd, 3rd order) to identify non-linearity. Analysis will be done with triplicate sample using the mean of each for fitting. Where significant non-linearity is identified, experiments will either be repeated, or the linearity limit truncated to include the valid linear range. This will include quadruplicate measurement of samples at 6 different concentrations (4x6)
Limit of Quantitation | Through study completion - approximately 6 months
  The limit of quantitation (LoQ) is defined as the lowest concentration at which results show <=20% imprecision (CLSI EP17-A2). The LoQ will be determined as part of linearity using replicates of 4-6 to calculate the coefficient of variation at concentrations at or near the vendor claim.
Specificity | Through study completion - approximately 6 months
  Specificity refers to the ability of the analytical method to differentiate the analyte of interest from related or unrelated compounds. Studies typically focus on common drugs and interferences. These studies will include addition of substances known to interfere with the analyte of interest (hemolysis, icterus, lipemia, biotin, etc.). The vendor package inserts will be used to finalize the list of interferences and the CLSI EP07 guideline will be used to define the approach (recovery experiments in the presence of high concentrations of interfering substances).
Reference Intervals | Through study completion - approximately 6 months
  Reference intervals will either be validated against existing vendor defined cut points or established pending the findings of the method comparison studies. For either, 200 samples from healthy volunteers will be used. Depending on the distribution of the results, either parametric or non-parametric calculation of the 95% central confidence interval will be established. For HbA1c, the Canadian Diabetes Association guidelines have universally defined cut point, which requires that the assay show good agreement with the predicate method for usability

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McCudden, PhD,FCACB,FACB,NRCC-CC,DABC, Principal Investigator — Eastern Ontario Regional Laboratory Association.
Locations (1):
- Bio-Test Laboratory Inc., Nepean, Ontario, Canada